CLINICAL TRIAL: NCT03183726
Title: A Follow-up Study to Evaluate the Safety for the Patients With ALLO-ASC-DFU Treatment in Phase 1 Clinical Trial of ALLO-ASC-DFU-101
Brief Title: A Follow-up Study to Evaluate the Safety of ALLO-ASC-DFU in ALLO-ASC-DFU-101 Clinical Trial
Status: Completed | Type: Observational
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-ASC-DFU-102
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ALLO-ASC-DFU treatment: Subjects with ALLO-ASC-DFU treatment in phase 1 clinical trial of ALLO-ASC-DFU-101
  Interventions: Biological: ALLO-ASC-DFU

INTERVENTIONS:
Biological: ALLO-ASC-DFU — ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide an new option in treating a diabetic foot ulcer.
  This study is a follow-up study without intervention.
  Other Names: Allogenic adipose-derived mesenchymal stem cells

SUMMARY:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 1 clinical trial (ALLO-ASC-DFU-101) for 23 months.

DETAILED DESCRIPTION:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 1 clinical trial (ALLO-ASC-DFU-101) for 23 months.

ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a Diabetic Foot Ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are treated with ALLO-ASC-DFU sheet in phase 1 clinical trial of ALLO-ASC-DFU-101.
2. Subjects who are able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Subjects who are considered not suitable for the study by the principal investigator (For example, Subjects requiring surgical procedure on target site).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject is enrolled who are treated with ALLO-ASC-DFU sheet in phase 1 clinical trial of ALLO-ASC-DFU-101.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 24 months
  Evaluation of AE

SECONDARY OUTCOMES:
Wound size and depth measurement | 6, 12, 24 months
  Evaluation of the improvement of wound measured by size and depth, and examines the change for 23 months period

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-suk Suh, MD, PhD, Principal Investigator — Asan Medical Center

IPD SHARING:
Plan to Share IPD: No